CLINICAL TRIAL: NCT06746116
Title: A Phase IIIB Study to Evaluate the Use of Durvalumab in Combination With Platinum-based Chemotherapy Followed by Durvalumab With Olaparib as First-line Treatment in Patients With Newly Diagnosed pMMR Advanced or Recurrent Endometrial Cancer in Spain
Brief Title: A Study to Evaluate the Use of Durvalumab in Combination With Platinum-based Chemotherapy Followed by Durvalumab With Olaparib as First-line Treatment in Advanced or Recurrent Endometrial Cancer in Spain
Acronym: DUoENDE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9311L00001
Record Dates: First submitted 2024-11-28; First posted 2024-12-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced or Recurrent Endometrial Cancer
Keywords: Durvalumab; Olaparib; pMMR; Endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Phase IIIb, interventional, single arm, multicentre study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Durvalumab + Chemotherapy (chemotherapy phase) plus Durvalumab + Olaparib (maintenence phase)
  Interventions: Drug: Durvalumab + Chemotherapy phase; Drug: Durvalumab + Olaparib phase

INTERVENTIONS:
Drug: Durvalumab + Chemotherapy phase — Durvalumab (IV) with SoC (carboplatin + paclitaxel chemotherapy: patients should receive at least 4, but preferably 6 cycles) every three weeks.
  Other Names: Chemotherapy phase
Drug: Durvalumab + Olaparib phase — durvalumab (IV) with olaparib (tablets) every four weeks until progression.
  Other Names: Maintenance phase

SUMMARY:
This is a phase IIIb, interventional, single arm, multicentre study assessing the safety profile of durvalumab in combination with carboplatin-paclitaxel chemotherapy followed by durvalumab with olaparib as first-line treatment for patients with pMMR aEC as the primary endpoint.

The study will include approximately 85 patients distributed in approximately 20 sites in Spain.

The planned duration of patient recruitment is approximately 12 months. Each patient will be followed up from screening for 36 months, until end of study period, death, withdrawal from study or loss to follow-up; whichever occurs first.

Enrolment will be opened to all eligible patients treated with durvalumab in combination with carboplatin-paclitaxel chemotherapy followed by durvalumab with olaparib as first-line treatment for patients with pMMR aEC. In addition, adequate tumour tissue before study entry, stool and blood sample collected will be required for central analysis to monitor the status of relevant biomarkers.

DETAILED DESCRIPTION:
The purpose of this study is to describe the safety profile of durvalumab in combination with platinum-based chemotherapy followed by durvalumab with olaparib as first-line treatment for patients with pMMR advanced or recurrent endometrial cancer.

Study population: Approximately 85 eligible patients with newly diagnosed pMMR advanced or recurrent endometrial cancer (aEC) will be enrolled into the study distributed in approximately 20 sites in Spain.

Study details include:

* The recruitment period will be approximately 12 months.
* The study duration will be approximately 48 months (12 months recruitment period + 36 months treatment and follow-up).
* The median treatment duration will be approximately 13 months based on treatment duration for durvalumab + olaparib in DUO-E (22) (until objective radiological disease progression, unacceptable toxicity, consent withdrawal or death). Those patients in complete response will be allowed to discontinue durvalumab plus olaparib after completing 2 years in the maintenance phase.
* The analysis for the primary objective is planned to be conducted 12 months after LSI to allow all patients have had the opportunity for 12 months of follow up, and at the end of the follow-up of the last patient up to 36 months.
* The visit frequency will be:

oChemotherapy Phase: every 21 days (every cycle). oMaintenance Phase: every 28 days (every cycle)

Treatment:

* Durvalumab + Chemotherapy phase: Durvalumab (IV) with SoC (carboplatin + paclitaxel chemotherapy: patients should receive at least 4, but preferably 6 cycles) every three weeks.
* Durvalumab + Olaparib phase: durvalumab (IV) with olaparib (tablets) every four weeks until progression.

ELIGIBILITY:
INCLUSION CRITERIA

Disease characteristics 3. Histologically confirmed diagnosis of endometrial carcinoma (all histologies, including carcinosarcoma) with archival or recent biopsy available to send at study entry.

4. Only patients with pMMR tumors are allowed (mismatch repair status determined locally per current clinical practice).

5. Patients must have endometrial cancer in one of the following categories:

1. Newly diagnosed Stage III disease classified by FIGO 2023 with mesurable disease per RECIST 1.1 following surgery or diagnostic biopsy.
2. Newly diagnosed Stage IV disease classified by FIGO 2023. Patients with primary cytoreduction without residual disease are allowed.
3. Recurrence of disease where the potential for cure by surgery alone or in combination is poor.

   6. Naïve to first-line systemic anti-cancer treatment. For patients with recurrent disease, prior systemic anti-cancer treatment is allowed only if it was administered in the adjuvant setting (for patients with FIGO 2023 stage II, III or IVA) and there is at least 6 months from date of last dose of adjuvant systemic treatment to date of subsequent relapse.

   7.At least one, but ideally two FFPE tumour sample block must be available and must be suitable for NGS and IHC evaluation by central lab. Preferably from primary endometrial tumor, but also from metastatic site will be allowed if there is no primary tumor block available. Tumor tissue has to have no less than 30% tumoral cell and tumoral area size has to be no less than 0,5cm2.

   8.Eastern Cooperative Oncology Group (ECOG)/ World Health Organisation (WHO) performance status ≤ 2 at enrolment.

   Note: not more than 20% of patients with ECOG PS2 will be allowed; once this limit is met, additional enrolled patients must have PS <2.

   Reproductive status 9.Postmenopausal or evidence of nonchildbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of Cycle 1 Day 1 and confirmed prior to treatment on Cycle 1 Day 1. Women will be considered post- menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:
   * Women <50 years of age will be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments, and if they have LH and FSH levels in the post- menopausal range for the institution.
   * Women ≥50 years of age will be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago.
   * Women who are surgically sterile (ie, bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) are eligible.

   Organ function 10.Adequate organ and bone marrow function, defined as:
   * Haemoglobin ≥10.0 g/dL
   * Absolute neutrophil count (ANC) ≥1.5 × 109/L
   * Platelet count ≥100 × 109/L
   * Serum bilirubin ≤1.5 × the upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome, who will be allowed in consultation with their physician.
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN; for patients with hepatic metastases, ALT and AST ≤5 × ULN.

     11.Measured creatinine clearance (CrCL) >51 mL/min or calculated CrCL >51 mL/min as determined by Cockcroft-Gault (using actual body weight), a 24-hour urine test or another validated test as per local practice: Estimated CrCL = (140-age [years]) × weight (kg) × 0.85 (mL/min) 72 × serum creatinine (mg/dL)

   EXCLUSION CRITERIA

   Participants are excluded from the study if any of the following criteria apply:

   Medical history
   1. Any unresolved toxicity National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE version 5.0) Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria. Note:

      -Patients with Grade ≥2 neuropathy may be included only after consultation with the study physician.

      -Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or olaparib may be included only after consultation with the study physician.
   2. Uterine sarcomas will not be allowed.
   3. Major surgical procedure (as defined by the investigator) within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery. Note: Local surgery of isolated lesions for palliative intent is acceptable or diagnostic staging.
   4. History of allogenic organ transplantation.
   5. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation.
   6. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

      -Patients with vitiligo or alopecia.

      -Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.

      -Any chronic skin condition that does not require systemic therapy.

      -Patients without active disease in the last 5 years may be included but only after consultation with the study physician.

      -Patients with coeliac disease controlled by diet alone.
   7. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension (systolic blood pressure >160 mmHg; diastolic blood pressure >100 mmHg), unstable angina pectoris, cardiac arrhythmia, interstitial lung disease (ILD), serious chronic gastrointestinal conditions associated with diarrhoea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
   8. History of another primary malignancy except for:

      -Malignancy treated with curative intent and with no known active disease.

      -≥5 years before the first dose of IP and of low potential risk for recurrence.

      -Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
      * Adequately treated carcinoma in situ without evidence of disease.
   9. History of leptomeningeal carcinomatosis.
   10. Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have a magnetic resonance imaging (MRI) (preferred) or computed tomography (CT) each preferably with IV contrast of the brain prior to study entry.
   11. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischaemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation ≥500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
   12. History of active primary immunodeficiency.
   13. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive HBV surface antigen [HbsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HbsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
   14. Myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML) or with features suggestive of MDS/AML.

       Prior/concomitant therapy
   15. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
   16. Prior treatment with PARP inhibitors.
   17. Any prior exposure to immune-mediated therapy, including (but not limited to) other anti CTLA-4, anti-PD-1, anti-PD-L1, or anti-programmed-cell-death ligand 2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines.
   18. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable. Prior hormonal therapy for cancer treatment must be stopped at least 7 days prior to first dose of study treatment.
   19. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

       * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
       * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
       * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
   20. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.

       Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
   21. Concomitant use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg, ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks.
   22. Concomitant use of known strong (e.g., phenobarbital, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for phenobarbital and 3 weeks for other agents.

       Other exclusions
   23. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
   24. Unable to swallow orally administered medication.
   25. Any gastrointestinal disorder likely to interfere with absorption of the study medication.
   26. Pregnant or breastfeeding.
   27. Patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after last dose of study intervention or 6 months after the last dose of olaparib, whichever is later.
   28. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Adverse Events | Time from enrollment up to at least 90 days after last dose of study treatment
  Safety and tolerability will be evaluated in terms of Adverse Events (AEs), Serious AEs (SAEs), and immune-mediated AEs (imAEs)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From date of enrollment through to disease progression, death, withdrawn from study, or end of study (approximately 48 months)
  Defined as the time from the date of first dose of treatment until the date of objective disease progression or death (by any cause in the absence of progression). The measure of interest is the median PFS.
Objective Response Rate (ORR) | From date of enrollment through to disease progression, death, withdrawn from study, or end of study (approximately 48 months)
  Defined as the percentage of patients with a confirmed investigator-assessed response of CR or PR and will be based on a subset of all included patients with measurable disease at baseline per the site investigator.
Duration of Response (DoR) | From date of enrollment through to disease progression, death, withdrawn from study, or end of study (approximately 48 months)
  Defined as the time from the date of first documented response (which is subsequently confirmed) until date of documented progression or death in the absence of disease progression.
Overall Survival (OS) | From date of enrollment through to disease progression, death, withdrawn from study, or end of study (approximately 48 months)
  Defined as the time from the date of first dose of treatment2 until death from any cause.
Change in EORTC QLQ-C30 score | From date of enrollment through to disease progression, death, withdrawn from study, or end of study (approximately 48 months)
  Change from baseline (enrollment) in EORTC QLQ-C30 score every 12 weeks until end of treatment or disease progression.
Change in EORTC QLQ-EN24 score | From date of enrollment through to disease progression, death, withdrawn from study, or end of study (approximately 48 months)
  Change from baseline (enrollment) in EORTC QLQ-EN24 score every 12 weeks until end of treatment or disease progression.
Clinically meaningful deterioration | From date of enrollment through to disease progression, death, withdrawn from study, or end of study (approximately 48 months)
  Percentage of patients having absolute change in EORTC-QLQ-C30 and EORTC-QLQ-EN24 score from baseline of ≥10 at 6, 12, 24 and 36 months after LSI.

CONTACTS AND LOCATIONS:
Locations (19):
- Spain (19):
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, El Palmar
  - Research Site, Girona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Salamanca
  - Research Site, San Sebastián
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Vigo
  - Research Site, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/